CLINICAL TRIAL: NCT02665507
Title: Evaluation of the Efficacy of Light Therapy for the Treatment of Back Pain in Pilots
Brief Title: Light Therapy for the Treatment of Back Pain in Pilots (LLL&Pilots)
Acronym: LLL&Pilots
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Hebrew University of Jerusalem (Other)
Responsible Party: Principal Investigator, Lilach Gavish, Study Director, Hebrew University of Jerusalem
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 0630-15-HMO
Record Dates: First submitted 2016-01-24; First posted 2016-01-27 (Estimated); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Back Pain
Keywords: Photobiomodulation; Aviation
MeSH Terms: conditions — Back Pain | interventions — Lasers

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- LLLI (Active Comparator): Subjects from this group will receive 6 biweekly physiotherapy treatment and in addition LLLI (low level laser irradiation) treatment performed with Gallium-Aluminium-Arsenide 808 nm laser ( GaAlAs 808nm laser ).
  Interventions: Device: GaAlAs 808nm laser
- Sham (Sham Comparator): Subjects from this group will receive 6 biweekly physiotherapy treatment and in addition sham LLLI treatment
  Interventions: Device: Sham

INTERVENTIONS:
Device: GaAlAs 808nm laser — Hand held superpulsed GaAlAs 808 nm LLLI
  Arms: LLLI
Device: Sham — Hand held laser that emits no LLLI
  Arms: Sham

SUMMARY:
Back pain is a common complaint among pilots. Current treatments include physiotherapy and chiropractic manipulations. Low-level laser irradiation (LLLI) in the visible to near-infrared range was shown to reduce neck and low back pain.

The purpose of the study is to evaluate the efficacy of Light Therapy for treatment of back pain in pilots.

DETAILED DESCRIPTION:
Background: Lumbar spine disorders are common conditions in pilots of various aircraft with etiology related to sub-optimal ergonomics, exposure to G-forces, the weight of the head gear and exposure to extensive vibrations. Current treatments include physiotherapy and chiropractic manipulations. Low-level laser irradiation (LLLI) is a non-ionizing, non-thermal irradiation within the visible to near infrared range of the light spectrum. LLLI has been used widely for alleviation of pain in inflammatory processes and acceleration of wound healing. A variety of clinical studies show that LLLT in the near infrared range may be useful in the treatment of back pain.

Objective: To evaluate the efficacy of Light Therapy for treatment of back pain in pilots.

Study design: Prospective, randomized, controlled double blind. Volunteers will receive biweekly physiotherapy treatment for 3 weeks. In addition to the physiotherapy treatment, half the volunteers will receive light therapy and half sham irradiation. Study evaluations will include physical examination by an orthopedic surgeon, subjective pain level by visual analogue scale, validated low back functional questionnaires, a generic functional questionnaire, and patient satisfaction scores. Volunteers will be invited for evaluations at 1 and 3 months after the final treatment.

ELIGIBILITY:
Inclusion Criteria:

* Pilot (current)
* Level of pain - moderate to severe low back pain (≥40 on the pain VAS)

Exclusion Criteria:

* Low back pain due to non-traumatic etiological causes (infection, tumor, osteoporosis, ankylosing spondylitis, fracture, inflammatory process, cauda equinal syndrome).
* Pregnant
* Recent (up to 1 year) history of trauma
* Current chronic pain other than low back pain
* Physical disability that prevents the patient to lie down/get up

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2024-05-03 (Actual); Study Completion 2024-07-03 (Actual)

PRIMARY OUTCOMES:
Time to reach minimal important change in pain level by visual analog scale (VAS) | within 4 months

SECONDARY OUTCOMES:
Change in pain level by VAS after 3 weeks compared to baseline (before treatment) | 3 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Lilach Gavish, PhD, Study Director — Hebrew University of Jerusalem; Yair Barzilay, MD, Principal Investigator — Shaare Zedek Medical Center
Locations (1):
- Aviation Medicine Unit, Ramat Gan, Israel

IPD SHARING:
Plan to Share IPD: No